CLINICAL TRIAL: NCT05245136
Title: Augsburg Longitudinal Plasma Study (ALPS) to Study Liquid Biopsy (LBx) as a Tool for Diagnostic Support, Assessment of Disease Progression, and Identification of Mutations During Disease Course in Patients With Solid Neoplasms Receiving Palliative Treatment
Brief Title: Augsburg Longitudinal Plasma Study for the Evaluation of Liquid Biopsy as Diagnostic Tool.
Acronym: ALPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: N67
Record Dates: First submitted 2021-11-08; First posted 2022-02-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Characteristics Disease; Metastatic Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained, with potential for extraction of DNA from at least one of the types of samples retained (FFPE-tissue, whole blood, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational trial of patients with metastatic cancer of various entities which aims at both clarifying the significance of liquid biopsy and establishing a foundation for translational research.

DETAILED DESCRIPTION:
ALPS is a prospective observational trial to assess liquid biopsy as diagnostic tool in patients with various metastatic neoplasms. Liquid biopsy will be correlated not only with the tissue biopsy, but also to imaging modalities and classical tumor markers. In addition, the study aims to investigate clonal heterogeneity and evolution of different cancers during patient treatment courses. A third aspect of the study is to survey and assess patients' knowledge about biomarkers and personalized medicine in general and about liquid biopsy as a new diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Histopathologically confirmed metastatic or locally advanced cancer
* No curative treatment options, except for germ cell tumors
* Written Agreement to be followed up at Augsburg University Medical Center
* Signed written informed consent for the Biobank Augsburg (Biobank-A)
* Willing to undergo treatment according to standard of care
* Availability or anticipated availability of tumor tissue at time point of inclusion
* Anticipated life expectancy of at least 3 months at time point of trial inclusion

Exclusion Criteria:

* Psychological condition that would preclude informed consent
* Additional tumor treatment between acquisition of tumor tissue and trial inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of patients with diagnosis of metastatic cancer at the University Hospital Augsburg.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of tumor mutations between tissue biopsy (TBx) and liquid biopsy (LBx) at diagnosis | through study completion, an average of 3 years
  Correlation of tumor mutations between TBx and LBx at diagnosis with TBx as reference method based on PPA (positive percent agreement) and NPA (negative percent agreement)
Concordance between TBx and LBx at disease progression | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Concordance between TBx and LBx at disease progression with TBx as reference method based on PPA (positive percent agreement) and NPA (negative percent agreement)

SECONDARY OUTCOMES:
Investigation of tumor heterogeneity as a prognostic marker | through study completion, an average of 3 years
  Correlation of known and potential oncogenic drivers with imaging modalities based on morphological therapeutic response: ORR in classical entities and pools of tumor entities with ≥ 40 patient sample size
Correlation of known and potential oncogenic drivers in LBx with DCR | through study completion, an average of 3 years
  Correlation of known and potential oncogenic drivers with imaging modalities based on morphological therapeutic response: DCR in classical entities and pools of tumor entities with ≥ 40 patient sample size
Correlation of known and potential oncogenic drivers in LBx with OS | through study completion, an average of 3 years
  Correlation of presence of known and potential oncogenic drivers in LBx with OS per classical tumor entities and pools of tumor entities with ≥ 100 patient sample size
Role of a single numeric value (Shannon-Heterogeneity Index) at diagnosis as a surrogate marker for tumor heterogeneity | through study completion, an average of 3 years
  to evaluate the role of a single numeric value (Shannon-Heterogeneity Index) at diagnosis as a surrogate marker for tumor heterogeneity

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Schmutz, MD, Principal Investigator — UH Augsburg
Locations (1):
- University Hospital Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No